CLINICAL TRIAL: NCT05112289
Title: White Matter Hyperintensities in Migraine: A Multi-modal Imaging Project to Classify Disease Pathology
Brief Title: A Study to Evaluate White Matter Hyperintensities in Migraine
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Catherine (Cat) Chong, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-006203
Record Dates: First submitted 2021-10-12; First posted 2021-11-08 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Migraine; Small Vessel Ischemic Disease; Multiple Sclerosis
MeSH Terms: conditions — Migraine Disorders; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Migraine cohort (Other): Women with migraine and presence of white matter hyperintensities (WMH) on clinical magnetic resonance imaging (MRI) will have brain neuroimaging.
  Interventions: Diagnostic Test: Brain Neuroimaging
- Small vessel ischemic (SVI) disease cohort (Other): Women diagnosed with SVI disease and presence of white matter hyperintensities (WMH) on clinical magnetic resonance imaging (MRI) will have brain neuroimaging.
  Interventions: Diagnostic Test: Brain Neuroimaging
- Multiple sclerosis (MS) cohort (Other): Women diagnosed with MS and presence of white matter hyperintensities (WMH) on clinical magnetic resonance imaging (MRI) will have brain neuroimaging.
  Interventions: Diagnostic Test: Brain Neuroimaging

INTERVENTIONS:
Diagnostic Test: Brain Neuroimaging — Non-invasive magnetic resonance imaging sequences will investigate metabolic signatures unique to migraine WMH. Imaging data will be used for development of artificial intelligence (AI) algorithms to classify the cause of WMHs.

SUMMARY:
The purpose of this research is to better understand brain white matter hyperintensities (WMH) in women with migraines

ELIGIBILITY:
Inclusion Criteria - Migraine (N=20):

* Female only.
* Ages 20-45 years.
* Presence of WMH on MRI.

Exclusion Criteria:

* History of SVI and/or history of MS or other neurological disease other than migraine.
* History of cancer or organ transplantation.
* Contraindication to MRI.
* Pregnancy.
* History of abnormal brain MRI other than WMH.
* Subjects not willing to comply with the study procedures will be removed from the study.

Inclusion Criteria - SVI disease (n=10):

* Female only
* Ages > 60 years.
* Presence of WMH on MRI.

Exclusion Criteria:

* History of migraine and/or history of MS or other neurological disease other than SVI.
* History of cancer or organ transplantation.
* History of abnormal brain MRI other than WMH.
* Pregnancy.
* History of abnormal brain MRI other than WMH.
* Subjects not willing to comply with the study procedures will be removed from the study.

Inclusion Criteria - MS (n=10):

* Female only.
* Ages 20-45.
* Presence of WMH on MRI.

Exclusion Criteria:

* History of migraine and/or history of SVI or other neurological disease other than MS.
* History of cancer or organ transplantation.
* History of abnormal brain MRI other than WMH.
* Pregnancy.
* History of abnormal brain MRI other than WMH.
* Subjects not willing to comply with the study procedures will be removed from the study.

Ages: 20 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
WMH imaging disease parameters | 3 months
  Radiological MRI assessment of WMH in migraine

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Chong, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No